CLINICAL TRIAL: NCT00535093
Title: A Comparison of Available Rapid Streptococcus A Tests in Community Clinics in Israel: Accuracy, Ease of Use and Acceptability.
Brief Title: An Assessment of Rapid Streptococcal Tests in Community Clinics in Israel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Collaborators: Dept of Family Medicine, Faculty of Medicine, Hebrew University, Jerusalem, Israel (Other)
Responsible Party: Ian MiskinMD, Clalit Health Services Jerusalem Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HT4152
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2009-09

CONDITIONS: Pharyngitis; Streptococcus Pyogenes Infection; Streptococcus Pyogenes Identification
Keywords: Pharyngitis; Community infections; Rapid Testing; Group A Streptococcus
MeSH Terms: conditions — Pharyngitis; Streptococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (No Intervention): All patients fulfilling inclusion criteria will be evaluated for GAS infection using both a rapid streptococcus test and also a standard throat culture
  Interventions: Device: rapid streptococcal testing

INTERVENTIONS:
Device: rapid streptococcal testing — Each patient will have both RST and standard throat culture performed. Final diagnosis and treatment will be determined by throat culture

SUMMARY:
There is a large over-use of antibiotics in family medicine, especially in upper respiratory tract infections.

This study is designed to determine if the use of rapid Streptococcal tests in primary care clinics can lower the rate of antibiotic use while not missing bacterial infections.

DETAILED DESCRIPTION:
Pharyngitis is a clinical diagnosis which requires antibiotic treatment only if caused by group A Streptococcus (GAS).

However, it is impossible to identify by clinical signs alone those patients whose symptoms are caused by this pathogen.

Diagnosis demands a throat culture, which requires at least 24 hours to rule in infection and 48 hours to rule it out.

Rapid Streptococcal tests (RST) based on antigen identification have been in use for over 10 years. These allow determination of the presence of GAS within 10 minutes using tests designed for point of care use.

While the specificity of these tests is generally reported as high (90-95%), the sensitivity is quoted at between 60% and 90% , depending on author affiliation, place of testing and type of test.

Various protocols have been put forward, these combine clinical signs (Centor criteria) with RST or throat cultures in order to lower antibiotic over-use.

These protocols are often under-used by primary physicians, even when RSTs are available.

Clalit health services, the largest HMO in Israel, has decided to evaluate all the RSTs available in the country in community clinic settings in order to determine the feasibility of adopting these tests to improve clinical care.

The sensitivity, specificity and ease-of-use will be assessed in 25 clinics in various settings (urban and rural). Gold standard will be a standard throat culture processed in the district laboratory.

The effect of point-of-care testing will be estimated by requiring physicians to decide on antibiotic use before receiving the result of the RST. (They will be free to change this decision after the test).

Clinics were selected by number of throat cultures sent in previous years. The number of patients was determined using the positivity rates of 2005. The results of this study will enable us to estimate the benefit and cost of adopting RSTs, and to determine in which situations they will be most efficacious.

ELIGIBILITY:
Inclusion Criteria:

* sore throat
* at least two Centor criteria:
* fever > 38 deg C or history of fever
* enlarged cervical lymph nodes
* tonsillar exudate
* lack of cough
* age 3-14 years

Exclusion Criteria:

* antibiotic treatment in preceding 7 days
* no informed consent

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7000 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
sensitivity of RST specificity of RST | 3-4 months

SECONDARY OUTCOMES:
ease of use effect on antibacterial prescribing | 3-4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ian N Miskin, MD, Principal Investigator — Clalit Health Services, Jerusalem district
Locations (1):
- Clalit Health Services, Jerusalem, Israel

REFERENCES:
- [Background] Humair JP, Revaz SA, Bovier P, Stalder H. Management of acute pharyngitis in adults: reliability of rapid streptococcal tests and clinical findings. Arch Intern Med. 2006 Mar 27;166(6):640-4. doi: 10.1001/archinte.166.6.640. PMID 16567603
- [Background] Gieseker KE, Mackenzie T, Roe MH, Todd JK. Comparison of two rapid Streptococcus pyogenes diagnostic tests with a rigorous culture standard. Pediatr Infect Dis J. 2002 Oct;21(10):922-7. doi: 10.1097/00006454-200210000-00007. PMID 12394813
- [Background] McIsaac WJ, Kellner JD, Aufricht P, Vanjaka A, Low DE. Empirical validation of guidelines for the management of pharyngitis in children and adults. JAMA. 2004 Apr 7;291(13):1587-95. doi: 10.1001/jama.291.13.1587. PMID 15069046
- [Background] Bisno AL, Gerber MA, Gwaltney JM Jr, Kaplan EL, Schwartz RH; Infectious Diseases Society of America. Practice guidelines for the diagnosis and management of group A streptococcal pharyngitis. Infectious Diseases Society of America. Clin Infect Dis. 2002 Jul 15;35(2):113-25. doi: 10.1086/340949. No abstract available. PMID 12087516
- [Background] Linder JA, Chan JC, Bates DW. Evaluation and treatment of pharyngitis in primary care practice: the difference between guidelines is largely academic. Arch Intern Med. 2006 Jul 10;166(13):1374-9. doi: 10.1001/archinte.166.13.1374. PMID 16832002
- [Background] Ebell MH, Smith MA, Barry HC, Ives K, Carey M. The rational clinical examination. Does this patient have strep throat? JAMA. 2000 Dec 13;284(22):2912-8. doi: 10.1001/jama.284.22.2912. PMID 11147989
- [Background] Linder JA, Bates DW, Lee GM, Finkelstein JA. Antibiotic treatment of children with sore throat. JAMA. 2005 Nov 9;294(18):2315-22. doi: 10.1001/jama.294.18.2315. PMID 16278359